CLINICAL TRIAL: NCT03564132
Title: A Randomized, Double-Blind, Placebo-Controlled Trial Evaluating the Efficacy and Safety of Yi-Gan San in Children and Adolescents With Tourette's Disorder
Brief Title: Evaluating the Efficacy and Safety of Yi-Gan San in Children and Adolescents With Tourette's Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMUH106-REC2-148
Record Dates: First submitted 2018-06-11; First posted 2018-06-20 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Tourette Disorder; Tic Disorders
Keywords: Yigansan; YGTSS
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yigansan (Experimental): 2.5g of Yigansan granules by mouth, three times a day for 4 weeks
  Interventions: Drug: Yigansan
- Placebo (Placebo Comparator): 2.5g of Placebo(contained one-tenth Yigansan) granules by mouth, three times a day for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Yigansan — Yigansan granules
  Other Names: YGS
  Arms: Yigansan
Drug: Placebo — One-tenth concentration of Yigansan manufactured to mimic Yigansan granules
  Other Names: Placebo (for Yigansan)
  Arms: Placebo

SUMMARY:
Yigansan was used in Ming dynasty by Xue Kai as a remedy for restlessness and agitation in children. We expect that the total YGTSS scores of Yigansan-treated subjects will be significantly reduced compared to that of placebo-treated subjects.

DETAILED DESCRIPTION:
Tourette's disorder (TD) is a chronic, childhood-onset neuropsychiatric disorder. It is characterized by multiple motor and vocal tics, including involuntary or semivoluntary, sudden, brief, intermittent, repetitive movements or sounds. Yigansan was used in several clinical trials, like dementia, pervasive developmental disorder, schizophrenia and Huntington's disease, with good results. So the investigators choose Yigansan as a Chinese medicine formula in this study. After the participants signed the consent form, they have to stop taking any Chinese medicine or western medicine for treating Tourette's disorder for two weeks and then are randomly assigned to Yigansan group or placebo group. Our hypothesis is that Yigansan will be expected to improve motor tics and vocal tics, and YGTSS scores will decrease after 4-weeks treatments; secondary outcomes are measured by CGI-TS (Clinical Global Impression-Tourette Syndrome) scale and GTS-QOL (The Gilles de la Tourette syndrome-quality of life scale), and the investigators will also proceed the basic research of metabolomics and biochemistry(GOT、GPT、BUN、Creatinine、K+). In order to ensure the relationship of Tourette's disorder and allergic rhinitis, the investigators will detect IgE. Besides, the investigators will collect blood and urine from every child or adolescent when a participant visits our clinic at week 0 and week 4. In order to find these biomarkers related to TD, the investigators will use ELISA kits to detect and quantitate significantly changeable concentration of cytokines associated with YGTSS scores. In addition to specific cytokine targets, the investigators will also find these metabolites involved in TD between two groups before and after taking YGS. The serum and urine samples will be prepared and subjected to LC-MS/MS analysis. In summary of the experimental designs and expected results, the therapy and background information will be more clarified on the therapeutic efficacy and safety by Yigansan treatment for TD. Most importantly, this study will provide a kind of Chinese medicine formula to relieve such a disorder that most doctors feel difficult to treat.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is a male or female child or adolescent, 6 to 17 years of age (inclusive) at the time of signing the informed consent/assent.
2. The subject meets current DSM-V diagnostic criteria for Tourette's Disorder.
3. The subject has a total score of ≥ 20 on the YGTSS at Screening and Baseline (randomization).
4. Tic symptoms may cause impairment in the subject's normal routines, which include academic achievement, occupational functioning, social activities, and/or relationships.
5. Females of childbearing potential (defined by menarche and not having undergone surgical sterilization/hysterectomy) must have a negative urine pregnancy test (when visiting our clinic at week 0 and week 4).

Exclusion Criteria:

1. The subject presents with a clinical presentation and/or history that is consistent with another neurologic condition that may have accompanying abnormal movements. These include, but are not limited to:

   Transient Tic disorder/ Huntington's disease/ Parkinson's disease/ Sydenham's chorea/ Wilson's disease/ Mental retardation/ Pervasive developmental disorder/ Traumatic brain injury/ Stroke/ Restless Legs Syndrome
2. The subject has a history of schizophrenia, bipolar disorder, or other psychotic disorder.
3. Subjects who receive psychostimulants for the treatment of ADD/ADHD and who have developed and/or had exacerbations of the tic disorder after the initiation of stimulant treatment.
4. Subjects who ever participated in any Chinese medicine or western medicine trial within 30 days.
5. Subjects requiring cognitive-behavioral therapy (CBT) for Tourette's Disorder during the trial period.
6. The inability to swallow Chinese herbal medicine.
7. Female subjects who have been pregnant.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2018-06-16 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Week 4 in Yale Global Tic Severity Scale (YGTSS) total tic score (TTS) | Baseline to Week4
  Ratings are 5 different dimensions on a scale of 0 to 5 for motor and vocal tics each, including number, frequency, intensity, complexity, and interference. The scores of TTS are from 0 to 50 and the scores of impairment are also from 0 to 50. Summation of TTS and impairment are YGTSS scores which will be the primary outcome measure in this trial.

SECONDARY OUTCOMES:
Change in Clinical Global Impressions Scale-Tourette's Syndrome (CGI-TS) Score at Week 4 | Baseline to Week 4
  Response choices included: 0 = not assessed; 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill patients. The change score was obtained from CGI-TS improvement scale assessment: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse.
Mean change from Baseline to Endpoint (Week 4) in Total YGTSS Score | Baseline to Week 4
  The YGTSS is used to rate the severity of symptoms (on a scale of 0 to 5 for 5 different dimensions, including number, frequency, intensity, complexity, and interference) of motor and vocal tics, and an impairment ranking. The Total YGTSS score is the summation of the severity scores of motor and vocal tics and also the ranking of impairment (range of 0 to 100).
Response Rate | Week 4
  Clinical response is defined as > 25% improvement from baseline to Week 4 in YGTSS TTS between 2 groups or a CGI-TS Change score of 1 [very much improved] or 2 [much improved] at Week 4.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Hao Huang, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jankovic J. Tourette's syndrome. N Engl J Med. 2001 Oct 18;345(16):1184-92. doi: 10.1056/NEJMra010032. No abstract available. PMID 11642235
- [Background] Cohen SC, Leckman JF, Bloch MH. Clinical assessment of Tourette syndrome and tic disorders. Neurosci Biobehav Rev. 2013 Jul;37(6):997-1007. doi: 10.1016/j.neubiorev.2012.11.013. Epub 2012 Dec 1. PMID 23206664
- [Background] Wang S, Qi F, Li J, Zhao L, Li A. Effects of Chinese herbal medicine Ningdong granule on regulating dopamine (DA)/serotonin (5-TH) and gamma-amino butyric acid (GABA) in patients with Tourette syndrome. Biosci Trends. 2012 Aug;6(4):212-8. doi: 10.5582/bst.2012.v6.4.212. PMID 23006968
- [Background] Zhao L, Li AY, Lv H, Liu FY, Qi FH. Traditional Chinese medicine Ningdong granule: the beneficial effects in Tourette's disorder. J Int Med Res. 2010 Jan-Feb;38(1):169-75. doi: 10.1177/147323001003800119. PMID 20233526
- [Background] Kim YH, Son CG, Ku BC, Lee HW, Lim HS, Lee MS. Herbal medicines for treating tic disorders: a systematic review of randomised controlled trials. Chin Med. 2014 Feb 7;9(1):6. doi: 10.1186/1749-8546-9-6. PMID 24507013
- [Background] Wu M, Xiao GH, Zhang JM, Zhang X, Ma B, Wang SX, Zhou YB, Zhang JY. Clinical research into Qufeng Zhidong Recipe used to treat 31 children with tic disorder. J Tradit Chin Med. 2010 Sep;30(3):163-70. doi: 10.1016/s0254-6272(10)60034-9. PMID 21053620
- [Background] Chou IC, Lin HC, Lin CC, Sung FC, Kao CH. Tourette syndrome and risk of depression: a population-based cohort study in Taiwan. J Dev Behav Pediatr. 2013 Apr;34(3):181-5. doi: 10.1097/DBP.0b013e3182829f2b. PMID 23572168
- [Background] Zheng Y, Zhang ZJ, Han XM, Ding Y, Chen YY, Wang XF, Wei XW, Wang MJ, Cheng Y, Nie ZH, Zhao M, Zheng XX. A proprietary herbal medicine (5-Ling Granule) for Tourette syndrome: a randomized controlled trial. J Child Psychol Psychiatry. 2016 Jan;57(1):74-83. doi: 10.1111/jcpp.12432. Epub 2015 Jun 13. PMID 26072932
- [Background] Eddy CM, Rickards HE, Cavanna AE. Treatment strategies for tics in Tourette syndrome. Ther Adv Neurol Disord. 2011 Jan;4(1):25-45. doi: 10.1177/1756285610390261. PMID 21339906
- [Background] Takeyoshi K, Kurita M, Nishino S, Teranishi M, Numata Y, Sato T, Okubo Y. Yokukansan improves behavioral and psychological symptoms of dementia by suppressing dopaminergic function. Neuropsychiatr Dis Treat. 2016 Mar 15;12:641-9. doi: 10.2147/NDT.S99032. eCollection 2016. PMID 27042075
- [Background] Miyaoka T, Furuya M, Horiguchi J, Wake R, Hashioka S, Thoyama M, Murotani K, Mori N, Minabe Y, Iyo M, Ueno S, Ezoe S, Hoshino S, Seno H. Efficacy and safety of yokukansan in treatment-resistant schizophrenia: a randomized, multicenter, double-blind, placebo-controlled trial. Evid Based Complement Alternat Med. 2015;2015:201592. doi: 10.1155/2015/201592. Epub 2015 Apr 14. PMID 25954314
- [Background] Miyaoka T, Furuya M, Horiguchi J, Wake R, Hashioka S, Tohyama M, Mori N, Minabe Y, Iyo M, Ueno S, Ezoe S, Murotani K, Hoshino S, Seno H. Efficacy and safety of yokukansan in treatment-resistant schizophrenia: a randomized, double-blind, placebo-controlled trial (a Positive and Negative Syndrome Scale, five-factor analysis). Psychopharmacology (Berl). 2015 Jan;232(1):155-64. doi: 10.1007/s00213-014-3645-8. Epub 2014 Jun 13. PMID 24923986